CLINICAL TRIAL: NCT05677737
Title: The Effect of Educatıon Gıven to Women on Breast Cancer Health Belıefs and Screenıng Behavıors,Randomized Controlled Trial
Brief Title: Women on Breast Cancer Health Belıefs and Screenıng Behavıors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, NİHAN TÜRKOĞLU, Assist Prof., Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: nihan25
Record Dates: First submitted 2022-12-29; First posted 2023-01-10 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer Female
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): In the study, the women in the experimental group will be trained every two weeks for 6 weeks.
  Interventions: Other: Education
- Control (No Intervention): No intervention will be applied to the control group.

INTERVENTIONS:
Other: Education — Educational program; It will be applied to the individuals in the experimental group for an average of 40 minutes in a time period they are suitable through the online platform prepared for the individuals in the experimental group in a three-month period. The literature will be scanned and appropriate educational materials will be created, and videos will be used to support education.
  Educational program During the first interview, the individuals in the experimental group will be introduced to the online platform, their entrance will be provided, they will be informed about how to follow the trainings, and sample applications will be made.
  Six main topics will be covered in the training program and will be completed every two weeks in three months.
  Arms: Experimental

SUMMARY:
Method: It was conducted in a randomized controlled experimental type. The population of the study consisted of 2426 women over the age of 20 living in a family health center in Erzurum between October 2021 and September 2022. The sample of the study consisted of 252 women with 0.05 margin of error and 95% confidence level, according to the sample size calculation formula used in cases where the universe is known. Within the framework of the exclusion criteria of the study, 52 women were excluded from the study and 200 women were included in the randomization.

DETAILED DESCRIPTION:
Persons in the experimental group will be trained 6 times with an interval of 2 weeks via an online platform (zoom, etc.). No training will be given to the control group, and the post-test data will be collected by re-administering the two groups with the mid-test created via Google forms and containing the scales immediately after the training, and the "Health Belief Model Scale in Breast Cancer Screening" and "Breast Cancer Screening Beliefs Scale" two months later.

ELIGIBILITY:
Inclusion Criteria:

-Being over 18 years old

* Being literate,
* Computer can be used,
* Internet is accessible,
* Not getting breast cancer before,

Exclusion Criteria:

* Having received training on breast cancer before

  * Having a history of breast cancer in first degree relatives
  * Those who did not attend all of the online trainings in the experimental group

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-05-28 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Breast Cancer Screening Beliefs Scale | two week
  Breast Cancer Screening Beliefs Questionnaire: The scale was developed by Kwok et al. (2010) in 2010 to determine women's breast cancer screening beliefs. Turkish adaptation, reliability, and validity of the scale were performed by Türkoğlu and Sis Çelik in 2021. The scale has three sub scales including Attitudes towards General Health Checkups, Knowledge and Perceptions about Breast Cancer, and Perceived Barriers to Mammographic Screening. Cronbach's alpha internal coefficients were found to range between 0.76 and 0.87 in the sub-scales of the original scale. The scores to be obtained from the scale range between 0 and 100. Mean scores of 65 and over in the sub-scales indicate that screening beliefs increase positively, knowledge level increases, and barriers to mammography screening decrease.
Health Belief Model Scale in Breast Cancer Screening | Two week
  This policy was first established by Champion in 1984 in the Health Belief Model base building. The scale has 8 dimensions: sensitivity, caring, health motivation, BSE barriers, benefits, self-efficacy, mammography benefits and barriers. Necessary components were tested, with the scale's caring and health motivation being revised in 1993, refinement in 1999, and BSE benefits, barriers, and self-efficacy dimensions revised again in 1997 (Champion, 1993; Champion and Scott, 1997; Champion, 1999; Champion, 1984) . Turkish validity and reliability were performed by Gözüm and Aydın in 2004. The scale includes subsections of "sensitivity", "caring", "health motivation", "BSE benefits", "BSE barriers", "BSE self-efficacy". The scale is a Likert-type scale scored from 1 to 5. A score closer to 5 means that caring, health motivation, BSE benefits, BSE barriers and BSE self-efficacy are perceived to be high.

CONTACTS AND LOCATIONS:
Overall Officials: Aslı Sis Çelik, Assoc. Prof., Study Chair — Ataturk University
Locations (1):
- Ataturk Unıversity, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No